CLINICAL TRIAL: NCT05480917
Title: Value Based Healthcare in Psoriasis - IRIS Trial
Brief Title: Value Based Healthcare in Psoriasis
Acronym: IRIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Novartis (Industry); Janssen, LP (Industry); Vlerick Business School (Unknown); Scientific Research Foundation-Flanders (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ONZ-2022-0184
Record Dates: First submitted 2022-07-20; First posted 2022-07-29 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Psoriasis
Keywords: Value-based healthcare; Psoriasis; Value
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: The IRIS trial will be a prospective clinical trial in which patients attending the PsoPlus for the first time will be followed during a period of 1 year. The focus will lie on patients with no prior experience with PsoPlus. The study will run for 24 months, of which 12 months will serve as an inclusion period. Both outcomes (VOS) and costs will be collected. The VOS is normally measured on a biannual basis. For this trial these time points are called T0, T1, and T2. Additionally, screening for comorbidities is performed to account for the integrated way of working. Patient as well as disease characteristics are also captured in a standardized way. This is all considered to be standard of care within PsoPlus. Cost data is collected using TD-ABC over the full cycle of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IRIS (Other)
  Interventions: Other: Patients receiving PsoPlus care

INTERVENTIONS:
Other: Patients receiving PsoPlus care — As stated before, both outcomes (via VOS) and costs will be collected. Data on clinical outcomes, such as skin clearance, in the VOS will be collected during follow-up visits at our clinic. Outcomes which are assessed via a questionnaire will be collected using a specialized patient platform (PsoQuest). In addition, for this study the EuroQol 5 Dimensions 5 Level (EQ-5D-5L) questionnaire will need to be filled in. When consultations do not coincide with the time points, data will be collected by a study nurse on a study visit (at our department or the patient's home) and via PsoQuest. A 1 month period will be in place around the time point, meaning that the data can be collected 2 weeks beforehand or afterwards. Cost data will be collected using the TD-ABC approach over the full cycle of care.

SUMMARY:
Rationale:

Currently, the healthcare sector is under tremendous financial pressure, and many acknowledge that a dramatic shift is required as the current system is not sustainable. Furthermore, the quality of care that is delivered varies strongly. Several solutions have been proposed of which the conceptual framework known as value-based healthcare (VBHC) is further explored in this study for psoriasis. Psoriasis is a chronic inflammatory skin disease which is associated with high treatment costs.

Objective:

The objective of this study is to investigate the impact of using the VBHC framework for the management of psoriasis.

Study design:

The IRIS (value In psoRiasIS) study will be a prospective clinical trial in which new patients attending the psoriasis clinic (PsoPlus) of the Ghent University Hospital will be followed up during a period of 1 year.

Study population:

The study population consists of psoriasis patients attending the PsoPlus for the first time.

Main study parameters/endpoints:

The main outcome is to determine the value created for new psoriasis patients in PsoPlus over a period of 1 year. Thus, the main study parameters pertain to clinically and patient reported outcomes as well as the full cost for treating patients under the year of review, including referrals to other departments. Secondary outcomes are related to comorbidity control, individual outcomes and determining cost drivers. In addition, a bundled payment scheme should be determined as well as potential improvements in the treatment process.

DETAILED DESCRIPTION:
The healthcare sector is under tremendous financial pressure but an increase in healthcare spendings does not seem to equate to better health outcomes or quality of care. Therefore, a dramatic shift is required as the current system is not sustainable. Several solutions have been proposed of which the conceptual framework known as value-based healthcare (VBHC) is further explored in this study for psoriasis. Psoriasis is a chronic inflammatory skin disease with a high prevalence of 0.1% to 11%. It is associated with psoriatic arthritis and numerous other comorbidities such as hypertension, obesity and diabetes. Psoriasis also significantly impacts patients' quality of life. The cost associated with managing psoriasis and its comorbidities present a substantial economic burden.

VBHC is a widely known conceptual framework, proposed by Porter and Teisberg, aimed at tackling the ever rising healthcare costs and variation in quality of delivered care. The framework is formulated on the premise that the health care sector should strive to achieve greater value for its patients. Value is defined through an equation in which the achieved patient-relevant outcomes are divided by the costs needed to achieve these outcomes. Both measures of outcomes and costs are looked at for individual patients over the full cycle of care, from the initial consultation to their final consultation, including all other medical interventions for the treatment of the medical disease. Previously, for psoriasis, it was unknown which outcomes actually mattered to patients. Therefore, a value-based outcome set (VOS), consisting of outcomes that matter to psoriasis patients, was first developed. Time-driven activity-based costing (TD-ABC) is the proposed costing method to accurately measure costs within the VBHC framework. Furthermore, in keeping with the VBHC framework, having greater understanding and transparency of costs may help with moving the sector away from the current fee-for-service structure towards VBHC payment initiatives, for example bundled payments. Bundled payments represent a lump sum payment to hospitals for the reimbursement of an entire episode of care for a patient. The payment is allocated to all services and providers across the various care activities (inpatient, post-acute care etc.).

In VBHC, value is created by using integrated practice units (IPUs). An IPU is an organizational entity that connects multiple specialisms and functions around a medical condition, with a distinct organizational structure, with a coherent set of agreements/contracts, with the aim to maximize value, by delivering maximum (or "the best possible") healthcare outcome for patients against minimum possible costs. It includes the full range of medical expertise, technical skills and specialized facilities needed, whilst putting patient experience central, as well as the management and coordination of the IPU and its interfaces. An IPU represents a fundamental part of the implementation of VBHC. The investigators have set up an IPU in psoriasis called PsoPlus, referring to the added value they believe their approach brings to psoriasis management.

The objective of this study is to investigate the impact of using the VBHC framework for the management of psoriasis. The IRIS (value In psoRiasIS) study will be a prospective clinical trial in which new patients attending the PsoPlus will be followed up during a period of 1 year. Both the outcomes achieved and costs will be assessed during this year. Subsequently, the two will be connected by conducting a data envelopment analysis (DEA) which will result in a value score for each patient. Based on this score and the evolution of this score conclusions can be made about the characteristics of patients that appear to experience more value compared to the other patients and the evolution of this created value over time. Secondary outcomes are related to comorbidity control, individual outcomes and determining cost drivers. In addition, a bundled payment scheme should be determined as well as potential improvements in the treatment process. This project will serve as a pilot project for the Belgium healthcare system.

The VOS consists of 21 outcomes which are measured using 12 instruments, of which 8 are reported by the patient and 4 by the provider. The following outcomes are measured:

* Symptom control via Psoriasis Symptom Inventory (PSI)
* Confidence in care via Patient Benefit Index (PBI)
* Control of disease via Patient Benefit Index (PBI)
* Treatment efficacy via Treatment Satisfaction Questionnaire for Medication (TSQM)
* Treatment convenience via Treatment Satisfaction Questionnaire for Medication (TSQM)
* Complete clearance via Psoriasis Area Severity Index (PASI) and Body Surface Area (BSA)
* Almost complete clearance via Psoriasis Area Severity Index (PASI) and Body Surface Area (BSA)
* Communication with care professional via Shared Decision-Making Questionnaire 9 item (SDM-Q9)
* Daily activity via Dermatology Life Quality Index (DLQI)
* Emotional well-being via Dermatology Life Quality Index (DLQI)
* Intimate relationships via Dermatology Life Quality Index (DLQI)
* Social activity via Dermatology Life Quality Index (DLQI)
* Difficult location clearance via Yes/No question in the Belgian Treat-to-Target consensus (T2T)
* Treatment tolerability via Yes/No question in the Belgian Treat-to-Target consensus (T2T)
* Treatment sustainability via custom Yes/No question
* Time to clearance via custom Yes/No question
* Cost of care (patient) via custom Yes/No question
* Cost of care (societal) via custom Yes/No question
* Treatment safety via Common Terminology Criteria for Adverse Events (CTCAE) criteria
* Productivity via Work Productivity and Activity Impairment - Psoriasis (WPAI-PSO)
* Comorbidity control via screening

ELIGIBILITY:
Inclusion Criteria:

* Dermatologist reported diagnosis of psoriasis vulgaris
* New patients that have never visited our specialized psoriasis consultation PsoPlus

Exclusion Criteria:

* Patients unable to provide consent
* Patients who previously visited our specialized psoriasis consultation PsoPlus within the last 5 years
* Patients who previously visited our psoriasis expert within the last 5 years
* Patients with an uncertain diagnosis of psoriasis
* Patients with all other subtypes of psoriasis
* Patients who are unable to understand the tasks and questionnaires

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
To determine the value created over a 1 year period while managing psoriasis patients within PsoPlus | 1 year
  The created value will be considered as a reflection of the evolution of the value score (i.e. the weighted outputs (outcomes in VOS) divided by weighted inputs (costs)) obtained using DEA

SECONDARY OUTCOMES:
Outcomes | At 6 and 12 months
  Determine change from baseline in VOS (all outcomes) at 6 and 12 months For a description of the VOS, see Detailed Study Description. The EQ-5D-5L will also be measured.
Outcomes | At 6 and 12 months
  Determine the relationship between individual outcomes For a description of the VOS, see Detailed Study Description. The EQ-5D-5L will also be measured.
Outcomes | At 6 and 12 months
  Determine variables (e.g. age, disease severity, treatment) that contribute to outcome variability For a description of the VOS, see Detailed Study Description. The EQ-5D-5L will also be measured.
Costs | At 6 and 12 months
  Determine total costs at 6 and 12 months
Costs | At 6 and 12 months
  Determine variables (e.g. age, disease severity, treatment) that contribute to cost variability
Outcomes/costs For a description of the VOS, see Detailed Study Description. The EQ-5D-5L will also be measured. | At 6 and 12 months
  Create patient profiles, that reflect efficient (experience more value) and inefficient (experience less value) patients, using DEA For a description of the VOS, see Detailed Study Description.
Comorbidities | At 6 and 12 months
  Assess the comorbidity evolution at 6 and 12 months (e.g. improvement (significant decrease) of cholesterol serum level) For a description of the VOS, see Detailed Study Description. The EQ-5D-5L will also be measured.
Comorbidities | At 6 and 12 months
  Determine number of comorbidities controlled (treated and below cut-offs) at 6 and 12 months For a description of the VOS, see Detailed Study Description. The EQ-5D-5L will also be measured.
Comorbidities | At 12 months
  Determine number of referrals to other specialists regarding comorbidities For a description of the VOS, see Detailed Study Description. The EQ-5D-5L will also be measured.
Bundled payments | At 12 months
  Determine a potential bundled payment scheme for treating different subsets of psoriasis patients over a particular time horizon
Integrated Practice Unit | At 12 months
  Improve the current IPU from an operational perspective by analyzing the value scores

CONTACTS AND LOCATIONS:
Overall Officials: Jo Lambert, Prof., Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - University Hospital Ghent, Ghent, East-Flanders
  - University Hospital Ghent, Ghent

IPD SHARING:
Plan to Share IPD: No
There are no plans to share IPD with other researchers.

REFERENCES:
- [Derived] Borzee J, Cardoen B, Roodhooft F, Vyvey E, Lambert J. Understanding psoriasis care costs and the impact of comorbidities: a time-driven activity-based costing analysis in an integrated practice unit. BMJ Open. 2026 Jan 9;16(1):e102879. doi: 10.1136/bmjopen-2025-102879. PMID 41513412
- [Derived] Hilhorst N, Roman E, Borzee J, Deprez E, Hoorens I, Cardoen B, Roodhooft F, Lambert J. Value in psoriasis (IRIS) trial: implementing value-based healthcare in psoriasis management - a 1-year prospective clinical study to evaluate feasibility and value creation. BMJ Open. 2023 May 23;13(5):e067504. doi: 10.1136/bmjopen-2022-067504. PMID 37221023